CLINICAL TRIAL: NCT07001046
Title: Effect of Mobile App-Based Exercises on Diastasis Rectus Abdominis in Post-Cesarean Mothers: A Randomized Controlled Trial
Brief Title: Impact of Mobile App-Based Exercises on Rectus Diastasis in Women Undergoing Cesarean Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Lecturer of Physical Therapy for Women's Health, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mobile App-Based Exercises
Record Dates: First submitted 2024-07-27; First posted 2025-06-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-07

CONDITIONS: Diastasis Recti and Weakness of the Linea Alba
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba

STUDY DESIGN:
Intervention Model Description: Two-arms Randomized Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 20 first-time mothers participated in a mobile app-guided exercise program focusing on abdominal muscles. The app was downloaded during their initial visit to supplement their treatment, which they conducted at home three times a week for eight weeks. They also attended follow-up sessions once a week.
  Interventions: Other: Mobile app-directed exercise program
- Group B (Experimental): 20 first-time mothers participated in a specific abdominal exercise program that included static abdominal exercises, head lifts with posterior pelvic tilting, and progressive curl-up exercises. The exercises were performed for 30 minutes, three times a week, for eight weeks as part of a home routine, along with a weekly follow-up session.
  Interventions: Other: Traditional Abdominal Exercises

INTERVENTIONS:
Other: Mobile app-directed exercise program — The mobile app-guided exercise program initially asks the mother questions to collect information. These questions were about their motivation for exercise, the main exercise goal, and the area of focus in the exercise program
  Arms: Group A
Other: Traditional Abdominal Exercises — The traditional abdominal exercises program consisted of simple static abdominal exercises, graduated curl-ups, and corrected abdominal crunches with posterior pelvic tilting
  Arms: Group B

SUMMARY:
Diastasis recti abdominis, or rectus diastasis, is the separation of the two parts of the rectus abdominis muscle along the midline of the linea alba, without any visible defect in the fascia.

Diastasis recti abdominis is most frequent during pregnancy and postpartum especially, after cesarean birth.

DETAILED DESCRIPTION:
Cesarean births were linked to significant post-operative changes in the thickness of abdominal fasciae and muscles when compared to vaginal births and these changes may be involved in the higher rates of diastasis recti post-cesarean births.

Managing diastasis recti abdominis begins with its diagnosis, followed by targeted interventions.

Diagnosis usually involves manual palpation to estimate the gap between the rectus abdominis muscles along the tendinous sheet of the linea alba. Updated imaging techniques, such as magnetic resonance imaging (MRI) and ultrasound, are now more frequently used for diagnosis.

Treatment either surgical or conservative; emphasizes physical therapy and personalized exercise programs. This method targets strengthening specific core muscles, such as the transverse abdominis and the pelvic floor.

ELIGIBILITY:
Inclusion Criteria:

* First-time mothers who delivered by a cesarean birth
* Post-cesarean women between 25 and 35 years old
* Women with a Diastasis Recti of at least 1 cm separation above the umbilicus and at least 0.5 cm separation below the umbilicus

Exclusion Criteria:

* First-time mothers who delivered by a vaginal birth
* Multiparous mothers
* Those who have not a Diastasis Recti
* Mothers under 25 years old and those above 35 years old

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study targeted the mothers who have a diastasis recti after cesarean birth
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Inter-recti Separation | Assessment was done pre treatment sessions and immediately after 8 weeks of treatment sessions
  The distance between the medial borders of the rectus abdominis muscles measured in Centimeters (cm) by the diagnostic Ultrasound.

SECONDARY OUTCOMES:
Abdominal muscle strength | Assessment was done pre treatment sessions and immediately after 8 weeks of treatment sessions
  A manual muscle test was used to assess the strength of rectus abdominis and abdominal obliques measured as an ordinal scale by a grading system of:
  Grade 0: No movement and no palpable contractions are evident.
  * Grade 1: No movement is possible but a flicker of a muscle contraction may be palpated.
  * Grade 2: With the arms held outstretched in front of the trunk, the patient lifts the head and cervical spine off the plinth. The scapulae remain on the plinth.
  * Grade 3: With the arms held outstretched in front of the trunk, the patient lifts the inferior angles of the scapulae clear of the plinth.
  * Grade 4: With the arms positioned across the chest, the patient lifts the inferior angles of the scapulae clear of the plinth.
  * Grade 5: With the hands positioned beside the ears, the patient lifts the inferior angles of the scapulae clear of the plinth.
Girth measurements | Assessment was done pre treatment sessions and immediately after 8 weeks of treatment sessions
  A tape measure examined waist, Umbilical, and Hip circumferences in centimeters (cm).
Satisfaction level | Assessment was done immediately after 8 weeks of treatment sessions
  A Questionnaire was used to assess the level of patient satisfaction with each treatment (grade 0; non-satisfaction for those have less than 9-10 on the Measure Yourself Medical Outcome Profile (MYMOP), and 1; satisfaction for those who have 9-10 on the MYMOP.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, South Valley University, Qina, Qena Governorate, Egypt